CLINICAL TRIAL: NCT00911781
Title: Hemangioma Growth During the First 6 Months of Life
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Mayo Clinic (Other); Medical College of Wisconsin (Other)
Responsible Party: Sponsor
Other Study IDs: hemangioma photo study
Record Dates: First submitted 2009-05-29; First posted 2009-06-02 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-02

CONDITIONS: Hemangiomas of Infancy
Keywords: Infantile hemangioma
MeSH Terms: conditions — Hemangioma, Capillary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Infants with infantile hemangiomas
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — We are only asking for photographs from parents.

SUMMARY:
One of the most important and unique characteristics of infantile hemangiomas is their dramatic growth during early infancy. Most hemangiomas are either absent at birth or barely evident as a small scratch or bruise-like area. A recent study emphasized how early hemangioma growth occurs. In this study by 3 months of age, hemangiomas had reached 80% of their final size, and by 5 months of age, 80% had already stopped growing. Unfortunately the average age when most infants are seen by specialists is often at 5 months of age or later, a time when most growth is already completed.

Researchers at the University of California, San Francisco, the Medical College of Wisconsin, and at the Mayo Clinic are interested in studying hemangioma growth at even earlier ages, before 3 months of age, which is before most patients are ever seen by dermatologists or other specialists. For this study are requesting that parents of children older than 3 months of age with hemangiomas send us a series of photographs of their child which demonstrates this early growth. Ideally the photographs would show your child (including the area of the hemangioma of course) at weekly or every other week intervals up until age least 3 to 6 months of age. This will probably not be difficult if the hemangioma is on the face but we would be interested in other body locations as well, if available.

We are using these photographs to analyze early hemangioma growth patterns, to see if there is a period of especially rapid growth, and to help determine if there is a specific time before which specialty referral should occur. We are interested in all sizes of hemangiomas, from small to large. Of greatest importance is that the photos be at frequent intervals (every 1 to 2 weeks is ideal) and of sufficient quality to be able to evaluate the appearance of the hemangioma.

ELIGIBILITY:
Inclusion Criteria:

* Children older than 3 months of age who have or have had a diagnosis of an infantile hemangioma. The parents of these children will be able to provide us with frequent (weekly to biweekly) photographs of the patient's hemangioma(s) during the first 3-6 months of life.
* These hemangiomas must have a superficial component that can be seen. Parents must consent to the use of their child's photographs in this study.

Exclusion Criteria:

* Current age less than 3 months. Patient who do not have an infantile hemangioma (as determined by the investigators). Patients whose photographs are not of sufficient quality or frequency in order to be evaluated for this study.

Ages: 3 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients are being recruited from a national hemangioma support website (NOVA)and from community clinics atthe University of California, San Francisco. We hope to reach more interested parents through registering our protocol.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2009-02; Primary Completion 2011-05 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
hemangioma growth | up to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ilona J Frieden, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - University of California, San Francisco, San Francisco, California
  - Mayo Clinic, Rochester, Minnesota

REFERENCES:
- [Background] Chang LC, Haggstrom AN, Drolet BA, Baselga E, Chamlin SL, Garzon MC, Horii KA, Lucky AW, Mancini AJ, Metry DW, Nopper AJ, Frieden IJ; Hemangioma Investigator Group. Growth characteristics of infantile hemangiomas: implications for management. Pediatrics. 2008 Aug;122(2):360-7. doi: 10.1542/peds.2007-2767. PMID 18676554
- See also: Tollefson MM, Frieden IJ. Early growth of infantile hemangiomas: what parents' photographs tell us. Pediatrics. 2012 Aug;130(2):e314-20. doi: 10.1542/peds.2011-3683. Epub 2012 Jul 23. PubMed PMID: 22826568. — http://www.ncbi.nlm.nih.gov/pubmed?term=tollefson%20m%20and%20frieden%20i&report=docsum&format=text